CLINICAL TRIAL: NCT03810560
Title: Microbiological and Clinical Assessments of Erbium Chromium: YSGG Laser as an Adjunctive to Surgical Treatment of Chronic Periodontitis (Randomized Clinical Trial)
Brief Title: Erbium Chromium: YSGG Laser Effect on Surgical Treatment of Chronic Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: alaa (Other)
Responsible Party: Sponsor-Investigator, alaa, Teaching Assistant, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER16-30M
Record Dates: First submitted 2019-01-05; First posted 2019-01-18 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Generalized Chronic Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- open flap debridement (No Intervention): surgical treatment of periodontal pocket without any intervention
- laser device with open flap debridement (Active Comparator): surgical intervention associated with application of Erbium chromium: YSGG laser therapy
  Interventions: Device: laser device Er,Cr:YSGG laser

INTERVENTIONS:
Device: laser device Er,Cr:YSGG laser — laser device with open flap debridement
  Arms: laser device with open flap debridement

SUMMARY:
Microbiological and Clinical assessment of Er,Cr:YSGG laser in conjunction to open flap debridement (OFD) in treatment of chronic periodontitis through real time PCR assay for quantification of total bacterial load.

DETAILED DESCRIPTION:
Two groups are randomly allocated (random number generation) by Microsoft excel into two groups :

1. Group (1) Open Flap debridement (OFD) surgery after conventional periodontal therapy (Scaling &Curettage and root planing) combined by Er,Cr:YSGG Laser assisted pocket therapy (ELAPT) which will be applied to pocket epithelial lining and root surface.
2. Group (2) Open Flap debridement (OFD) surgery after conventional periodontal therapy (Scaling &Curettage and root planing) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients are diagnosed to have chronic periodontitis, having infrabony posterior periodontal pocket measuring 5 mm or more.
* female or male.
* 25 - 55 years.
* Medically controlled according to medical coding of review of systems .
* Patient without history of drug administration in last month .

Exclusion criteria:

* Tobacco smoking.
* Pregnancy.
* Patients not follow periodontal hygienic instructions.
* Patients under any medication that affect periodontal healing.
* The presence of any systemic disease that affect periodontal healing.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Clinical Assessment of Plaque index(PI) | 6 months
  Visual Analog Score for plaque for detection amount of plaque accumulation so assess patient oral hygiene.
  recording is based on both soft and mineralized debris. Each surface will have a score from 0 to 3. 0: no plaque
  1. plaque only detected by probe.
  2. Moderate deposits detected by naked eye.
  3. heavy deposits detected by naked eye.
Clinical Assessment of Gingival index(GI) to assess gingival inflammation. 0: normal gingiva. 1: mild inflammation . 2: moderate inflammation . 3: sever inflammation marked redness and edema and spontaneous bleeding. | 6 months
  Visual Analog Score for gingival inflammation
Clinical Assessment of Probing depth (PD). | 6 months
  measured by milli meters for detection of level of periodontal destruction.
Clinical Assessment of Clinical attachment level (CAL) . | 6 months
  measured by milli meters for detection of level of periodontal destruction.
Clinical Assessment of Gingival recession(GR) | 6 months
  measured by milli meters for detection of level of apical migration of gingival attachment.
Clinical Assessment of Modified sulcular bleeding index (MSBI) | 6 months
  Visual Analog Score of bleeding for detection of inflammatory status level. Modified Sulcus Bleeding Index(MSBI) 0 = No bleeding on bleeding.
  1. =pin pointed bleeding.
  2. = linear bleeding.
  3. = Heavy or profuse bleeding.

SECONDARY OUTCOMES:
Microbiological assessment through real time PCR assay for quantification of total bacterial load by universal probe and primer set (16sr RNA) | 3 months
  quantification of total bacterial load

IPD SHARING:
Plan to Share IPD: No